CLINICAL TRIAL: NCT02160340
Title: Phase 1 Study of Optical Coherence Tomography Images to Identify the Prevalence of Vitreomacular Adhesion and Associated Maculopathies
Brief Title: Prevalence of Vitreomacular Adhesion in Patients 40 Years and Older
Acronym: VAST
Status: Completed | Type: Observational
Sponsor: Nova Southeastern University (Other)
Collaborators: ThromboGenics (Industry); Carl Zeiss Meditec, Inc. (Industry); Optovue (Industry)
Responsible Party: Sponsor
Other Study IDs: 11221319Exp
Record Dates: First submitted 2014-06-02; First posted 2014-06-10 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Vitreomacular Adhesion
Keywords: Posterior Vitreous Detachment; Vitreomacular Traction; Vitreous
MeSH Terms: conditions — Vitreous Detachment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vitreomacular adhesion: Male or female subjects aged over 40 years with vitreomacular adhesion

SUMMARY:
The purpose of this study is to evaluate the prevalence of vitreomacular adhesion (VMA) in patients 40 years and older using Spectral Domain Optical Coherence Tomography.

DETAILED DESCRIPTION:
As a function of age, liquefaction of the vitreous body results in separation of the vitreous cavity from the retina. This posterior vitreous separation may be incomplete, leading to areas of residual VMA. These adhesions can result in maculopathies such as vitreomacular traction syndrome, macular hole, epiretinal membrane, cystoid macular edema, diabetic macular edema, neovascularization in diabetic retinopathy and retinal vein occlusion, exudative age-related macular degeneration, and myopic traction maculopathy. VMA may lead to pathological sequelae due to the static and dynamic anteroposterior tractional forces to the surface of the macula. The resultant complication will depend on the size and strength of the traction, with smaller areas of adhesion leading to greater traction. Identifying the prevalence of vitreomacular adhesion and its associated complications will yield valuable, new epidemiologic data, leading to improved diagnosis and management of patients with this condition. The prevalence of vitreomacular adhesion in specific age groups has not been investigated.

ELIGIBILITY:
Inclusion Criteria: 40 years and older

* Clear media

Exclusion Criteria: Less than 40 years of age

* Prior history of vitreoretinal surgery or pharmacotherapy with intravitreal injection
* Dense media opacity

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from primary eye care clinics within academic settings, tertiary care clinics, and veterans administration medical centers.
Sampling Method: Probability Sample
Enrollment: 1584 (Actual)
Dates: Start 2014-05; Primary Completion 2016-01 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
What is the overall prevalence of Vitreomacular adhesion in the population 40 years and older? | Two years
  Prevalence will be measured using Spectral Domain Optical Coherence Tomography. Tomography scans will be evaluated for the presence or absence of vitreomacular adhesion.

SECONDARY OUTCOMES:
Is there is a significant correlation between VMA and various maculopathies including diabetic macular edema, retinal vascular occlusion, and age-related macular degeneration? | 2 years
  Spectral domain optical coherence tomography scans will be used to evaluate for the presence of isolated or concomitant vitreomacular adhesion.

OTHER OUTCOMES:
Is VMA more common in males or females? | 2 years
  The prevalence of VMA in both genders will be identified using Spectral Domain Optical Coherence Tomography and evaluated for statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Rodman, OD, MS, FAAO, Principal Investigator — Nova Southeastern University
Locations (18):
- United States (18):
  - Schaeffer Eye Center, Birmingham, Alabama
  - Leo Semes, Birmingham, Alabama
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - VA Greater Los Angeles Healthcare System, Sepulveda, California
  - Front Range Eye Associates, Broomfield, Colorado
  - Aran Eye Associates, Coral Gables, Florida
  - Nova Southeastern University, Fort Lauderdale, Florida
  - Retina Macula Specialists of Miami, Miami, Florida
  - Murray Ocular Oncology and Retina, Miami, Florida
  - Vitreous and Retina Consultants, Winter Haven, Florida
  - Clayton Eye Center, Morrow, Georgia
  - Indiana University College of Optometry, Indianapolis, Indiana
  - Grin Eyecare, Olathe, Kansas
  - Jones Eyecare, Albuquerque, New Mexico
  - Pacific University College of Optometry, Portland, Oregon
  - Larry Alexander, McKinney, Texas
  - Retina and Macula Specialists, Tacoma, Washington
  - Suburban Opticians, University Place, Washington